CLINICAL TRIAL: NCT05071807
Title: Cardiometabolic Effects of Including Pecans as a Snack to Improve Diet Quality: a Randomized Controlled Study
Brief Title: Cardiometabolic Effects of Pecans as a Snack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: American Pecan Council (Other)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PKE PECAN
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pecan Group (Active Comparator): Participants will consume their usual diet, but replace one snack with unsalted raw pecans incorporated as a snack
  Interventions: Drug: Pecans
- Usual Care Group (Active Comparator): Participants will consume their usual diet devoid of nuts
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Pecans — Participants will receive 2 oz of pecans daily to replace a typical snack and continue consuming their usual diet for 12 weeks.
  Arms: Pecan Group
Other: Usual Care — Participants will receive grocery vouchers and continue consuming their usual diet for 12 weeks.
  Arms: Usual Care Group

SUMMARY:
A randomized, 2-arm, parallel trial will be conducted to examine the effect of pecans on markers of peripheral vascular health, lipids and lipoproteins, blood pressure, and glycemic control.

DETAILED DESCRIPTION:
A randomized, 2-arm, parallel trial will be conducted to examine the effect of including 2 oz./day of pecans, as a snack, compared to a diet typically consumed by participants intake (devoid of nuts) on markers of peripheral vascular health, lipids and lipoproteins, blood pressure, and glycemic control. Participants will be randomized to pecans or control for 12-weeks. Outcome assessments will be measured at baseline and 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-40 kg/m2
* ≥ 1 criterion for metabolic syndrome (i.e., waist circumference ≥ 94 cm men or ≥ 80 cm women; triglycerides ≥150 mg/dL; HDL-cholesterol ≤ 40 mg/dL men or ≤ 50 mg/dL women; systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg; fasting plasma glucose ≥100 mg/dL) at screening

Exclusion Criteria:

* Current use of tobacco-containing products or (≤6 months) cessation
* Allergy/sensitivity/intolerance/dislike of study foods
* Women who are pregnant, lactating, planning to become pregnant or have given birth in the past year
* Individuals who have had a cardiovascular event (heart attack, revascularization, stroke), or have a history of heart failure, liver, kidney, autoimmune diseases or inflammatory conditions such as gastrointestinal disorders or rheumatoid arthritis.
* Type 1 or type 2 diabetes
* Unstable weight ≥10% body weight for 6 months prior to enrollment
* Systolic Blood pressure >160 mmHg for systolic pressure and/or diastolic blood pressure >/100 mmHg for diastolic pressure at screening
* Fasting blood glucose ≥126 mg/dL at screening
* Triglycerides ≥350 mg/dL at screening
* Taking any medications known to affect lipids, blood pressure, or blood glucose levels
* Diagnosed inflammatory conditions or taking prescribed , taking any chronic anti-inflammatory medications (>1 time per week over the past 3 months)
* Use of antibiotics within the prior 8 weeks
* Taking supplements (e.g., psyllium, fish oil, soy lecithin, and phytoestrogens) and botanicals known to affect study outcomes and not willing to cease for the duration of the study
* Individuals consuming >14 alcoholic drinks/week, and not willing to avoid alcohol consumption for 48 hours prior to test visit
* Pre-menopausal women who do not have a regular menstrual cycle of 25-35 days
* PI discretion

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Petersen, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hart TL, Kris-Etherton PM, Petersen KS. Nutrient Displacement Associated with Replacing Intake of Usual Snacks with Pecans: An Exploratory Analysis of a Randomized Controlled Trial. Curr Dev Nutr. 2025 Apr 9;9(5):107438. doi: 10.1016/j.cdnut.2025.107438. eCollection 2025 May. PMID 40386548
- [Derived] Hart TL, Kris-Etherton PM, Petersen KS. Pecan Intake Improves Lipoprotein Particle Concentrations Compared with Usual Intake in Adults at Increased Risk of Cardiometabolic Diseases: A Randomized Controlled Trial. J Nutr. 2025 May;155(5):1459-1465. doi: 10.1016/j.tjnut.2025.03.014. Epub 2025 Mar 18. PMID 40113170
- [Derived] Hart TL, Kris-Etherton PM, Petersen KS. Consuming pecans as a snack improves lipids/lipoproteins and diet quality compared with usual diet in adults at increased risk of cardiometabolic diseases: a randomized controlled trial. Am J Clin Nutr. 2025 Apr;121(4):769-778. doi: 10.1016/j.ajcnut.2025.01.024. Epub 2025 Jan 27. PMID 39880306

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pecan Group | Usual Care Group
Started | 69 | 69
Completed | 62 | 68
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Unrelated medical issues | 3 | 0
Not completed — Relocated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pecan Group | Usual Care Group | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12) | 46 (14) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 36 | 81
  Male | 24 | 33 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 138
Weight [Mean (Standard Deviation); unit: kg] | 84.3 (12.5) | 85.2 (14.3) | 84.8 (13.4)
Waist circumference [Mean (Standard Deviation); unit: cm] | 97.2 (8.8) | 98.8 (10.8) | 98.0 (9.9)
Pulse wave velocity [Mean (Standard Deviation); unit: m/s] | 7.1 (1.3) | 7.2 (1.2) | 7.2 (1.3)
Flow mediated dilation [Mean (Standard Deviation); unit: percent point change in arterial diamete] — FMD unit is percentage point change in brachial artery Flow Mediated Dilation (FMD). Higher values are associated with lower risk of cardiovascular events https://doi.org/10.1093/eurheartj/ehz350.
  percent point change in arterial diamete | 7.2 (4.0) | 6.1 (3.3) | 6.6 (3.7)
LDL-C [Mean (Standard Deviation); unit: mg/dL] | 118 (34) | 116 (28) | 117 (31)
HDL-C [Mean (Standard Deviation); unit: mmHg] | 54 (14) | 52 (13) | 53 (13.4)
Triglycerides [Mean (Standard Deviation); unit: mmHg] | 109 (67) | 116 (47) | 113 (58)
LDL subclasses [Mean (Standard Deviation); unit: nmol/L] — LDL particle size classifications are as follows: 22-25.5 nm is small, 25.6-26.5 nm medium, and 26.6-28.5 nm large. Typically, smaller LDL is associated with increased cardiovascular risk compared to larger.
  nmol/L
    Large | 373 (251) | 329 (194) | 351 (225)
    Medium | 366 (267) | 312 (255) | 339 (261)
    Small | 623 (435) | 698 (353) | 660 (396)
    Total LDL particle count | 1362 (399) | 1339 (339) | 1350 (396)
HDL subclasses [Mean (Standard Deviation); unit: µmol/L] — Size classifications of HDL subclasses are as follows: large (size 9.4-14.0 nm), medium (8.3-9.3 nm), and small (7.3-8.2 nm). Higher levels of large HDL may be inversely related to cardiovascular risk.
  µmol/L
    Large | 2.5 (1.7) | 2.3 (1.4) | 2.4 (1.6)
    Medium | 4.0 (1.8) | 4.4 (2.4) | 4.2 (2.1)
    Small | 14.2 (2.8) | 14.0 (3.4) | 14.1 (3.1)
    HDL total particle count | 20.7 (2.6) | 20.6 (2.9) | 20.7 (2.7)
Brachial blood pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 124 (15) | 125 (11) | 124 (13)
  Diastolic | 79 (8) | 79 (10) | 79 (9)
Central blood pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 114 (14) | 114 (14) | 114 (12)
  Diastolic | 79 (10) | 80 (8) | 80 (9)
Augmentation index @ 75bpm [Mean (Standard Deviation); unit: percentage of aortic pulse pressure] — Augmentation index is a measure of arterial stiffening that correlates with CVD risk. Higher augmentation index, used as a surrogate for wave reflection, is indicative of additional load on the left ventricle. Augmentation index is calculated as augmentation pressure/pulse pressure*100 to provide a percent. We utilized the Sphymocor Xcel for this measure. We used standardized augmentation index at 75 bpm for heart rate.
  percentage of aortic pulse pressure | 22 (11) | 21 (13) | 22 (12)
Plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 97 (7) | 98 (8) | 98 (7.4)
Serum insulin [Mean (Standard Deviation); unit: μIU/mL] | 9.4 (5.0) | 8.8 (3.5) | 9.1 (4.3)
HbA1C [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 5.5 (0.3) | 5.5 (0.3) | 5.5 (0.3)
Diet quality: Healthy Eating Index 2020 [Mean (Standard Deviation); unit: scores on a scale] — The Healthy Eating Index-2020 (HEI-2020) includes 13 components; 9 components are adequacy (i.e., consuming more results in a higher score), and 4 are moderation (i.e., consuming less results in a higher score) and measures adherence to the Dietary Guidelines for Americans 2020-2025. The simple HEI scoring algorithm per person was used with all reliable recalls from each timepoint to determine the HEI-2020 score for the timepoint. Scores range from 0 indicating no adherence to the dietary guidelines to 100 showing perfect adherence.
  scores on a scale | 57.2 (13.4) | 55.1 (10.7) | 56.1 (12.1)
Total Cholesterol concentration [Mean (Standard Deviation); unit: mg/dL] | 194 (39) | 190 (32) | 192 (36)

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation
Description: Measured by brachial ultrasound and expressed as percentage points of change in arterial diameter
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: percent point change in arterial diamete
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 67
percent point change in arterial diamete | 7.07 (0.35) | 7.25 (0.33)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; To detect a 1.2 percentage point (standard deviation 2.4; effect size 0.5) between-group difference in the change in FMD with 80% power (α=0.05), it was estimated that a sample size of 128 participants was needed (64 per group); Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and BMI (kg/m2); Mean Difference (Net) = 0.08, 95% CI 2-sided [-1.17 to 1.33]

2. Secondary Outcome: LDL-cholesterol Concentration
Description: Assessed from fasting blood draw expressed in mg/dL
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mg/dL | 110 (1.35) | 117 (1.26)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -7.2, 95% CI 2-sided [-12.3 to -2.1]

3. Secondary Outcome: HDL-cholesterol Concentration
Description: Assessed from fasting blood draw expressed in mg/dL
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mg/dL | 54 (0.47) | 53 (0.44)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = 1.1, 95% CI 2-sided [-0.8 to 2.9]

4. Secondary Outcome: Triglycerides
Description: Assessed from fasting blood draw expressed in mg/dL
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mg/dL | 97.7 [92.6 to 103] | 108 [103 to 114]
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -16.4, 95% CI 2-sided [-30.0 to -2.9]

5. Secondary Outcome: LDL Lipoprotein Subclasses
Description: Assessed from fasting blood draw expressed in nmol/L. Data were log transformed and back transformed to improve residual distribution; Measure Description: LDL particle size classifications are as follows: 22-25.5 nm is small, 25.6-26.5 nm medium, and 26.6-28.5 nm large. Typically, smaller LDL is associated with increased cardiovascular risk compared to larger.
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
nmol/L
  Large | 281 [249 to 317] | 252 [225 to 281]
  Total | 1248 [1216 to 1280] | 1304 [1273 to 1336]
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Total LDL particle mean difference; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -75.3, 95% CI 2-sided [-144 to -6.93]
Statistical Analysis 2: Comparison: Pecan Group vs Usual Care Group; For Large LDL particle subclass; Test type: Superiority; Regression, Linear; adjustment for the baseline value, age (years), sex (male or female) and body mass index (BMI) (kg/m2); Mean Difference (Net) = -27.9, 95% CI 2-sided [-69.3 to 13.4]

6. Secondary Outcome: HDL Lipoprotein Subclasses
Description: Assessed from fasting blood draw expressed in µmol/L; Measure Description: Size classifications of HDL subclasses are as follows: large (size 9.4-14.0 nm), medium (8.3-9.3 nm), and small (7.3-8.2 nm). Higher levels of large HDL may be inversely related to cardiovascular risk.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
μmol/L
  Medium | 4.1 (0.1) | 4.4 (0.1)
  Small | 14.1 (0.2) | 14.3 (0.2)
  Total | 21.0 (0.17) | 21.0 (0.16)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Results for total HDL particle count; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.56 to 0.75]
Statistical Analysis 2: Comparison: Pecan Group vs Usual Care Group; Results for Small HDL particles; Test type: Superiority; Adjusted for baseline value, age, sex, and BMI; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.75 to 0.80]
Statistical Analysis 3: Comparison: Pecan Group vs Usual Care Group; Results for Medium HDL; Test type: Superiority; Regression, Linear; Adjusted for baseline value, age, sex, and BMI; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.85 to 0.19]

7. Secondary Outcome: Brachial Systolic and Diastolic Blood Pressure
Description: Blood pressure measured assessed using a SphygmoCor Xcel (Atcor Medical)
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mmHg
  Systolic | 125 (0.81) | 125 (0.77)
  Diastolic | 79 (0.50) | 79 (0.47)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Results from brachial systolic blood pressure are reported below; Test type: Superiority; Regression, Linear; were adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-3.09 to 3.13]
Statistical Analysis 2: Comparison: Pecan Group vs Usual Care Group; Results for Brachial Diastolic Blood pressure; Test type: Superiority; Regression, Linear; Adjusted for baseline value, age, sex, BMI; Mean Difference (Net) = 0.20, 95% CI 2-sided [-1.67 to 2.07]

8. Secondary Outcome: Central Systolic and Diastolic Blood Pressure
Description: Blood pressure measured assessed using a SphygmoCor Xcel (Atcor Medical)
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mmHg
  Systolic | 114 (0.70) | 115 (0.69)
  Diastolic | 80 (0.50) | 80 (0.48)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Results for central systolic blood pressure; Test type: Superiority; Regression, Linear; Adjusted for baseline value, age, sex, BMI; Mean Difference (Net) = -0.48, 95% CI 2-sided [-3.24 to 2.28]
Statistical Analysis 2: Comparison: Pecan Group vs Usual Care Group; Results for central diastolic blood pressure; Test type: Superiority; Regression, Linear; Adjusted for baseline value, age, sex, BMI; Median Difference (Net) = 0.21, 95% CI 2-sided [-1.69 to 2.10]

9. Secondary Outcome: Carotid-femoral Pulse Wave Velocity
Description: A measure of arterial stiffness assessed using a SphygmoCor Xcel (Atcor Medical). Expressed in meters/second. Higher values indicate greater arterial stiffness
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
m/s | 7.1 (1.3) | 7.3 (1.3)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; were adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.26 to 0.24]

10. Secondary Outcome: Augmentation Index@75bpm
Description: A measure of arterial stiffness assessed using a SphygmoCor Xcel (Atcor Medical). Expressed as a percentage. A higher percentage value is indicative of greater arterial stiffness. Measure Description: Augmentation index is a measure of arterial stiffening that correlates with CVD risk. Higher augmentation index, used as a surrogate for wave reflection, is indicative of additional load on the left ventricle. Augmentation index is calculated as augmentation pressure/pulse pressure*100 to provide a percent. We utilized the Sphymocor Xcel for this measure. We used standardized augmentation index at 75 bpm for heart rate.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage of aortic pulse pressure
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
percentage of aortic pulse pressure | 21 (0.65) | 22 (0.65)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -1.65, 95% CI 2-sided [-4.25 to 0.95]

11. Secondary Outcome: Fasting Plasma Glucose Concentration
Description: Fasting blood glucose assessed by blood draw and expressed in mg/dL
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mg/dL | 97.7 (0.48) | 96.7 (0.45)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = 1.2, 95% CI 2-sided [-0.6 to 3.0]

12. Secondary Outcome: Serum Insulin Concentration
Description: Fasting serum insulin levels assessed by blood draw and expressed in micro IU/m
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: μIU/mL
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
μIU/mL | 8.42 [7.92 to 8.95] | 8.33 [7.87 to 8.83]
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.3 to 1.6]

13. Secondary Outcome: HbA1c
Description: HbA1c assessed in whole blood collected during fasting
Time Frame: 12-weeks
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
percentage of glycated hemoglobin | 5.53 (0.01) | 5.49 (0.01)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = 0.0, 95% CI 2-sided [0.0 to 0.1]

14. Secondary Outcome: Diet Quality: Healthy Eating Index 2020
Description: Diet quality measured by 24-hour recalls will be assessed using Health Eating Index 2020 (HEI-2020) scores range from 0-100 with 100 indicating perfect adherence to dietary guidelines and 0 indicating no adherence. The HEI-2020 includes 13 components; 9 components are adequacy (i.e., consuming more results in a higher score), and 4 are moderation (i.e., consuming less results in a higher score). The HEI-2020 was calculated with the Statistical Analysis System (SAS) code from the National Cancer Institute.
Time Frame: 12-weeks
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 65 | 67
scores on a scale | 60.8 (1.1) | 51.5 (1.0)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Mixed Models Analysis — When a significant group by time point interaction was detected, post hoc testing was conducted and the Tukey-Kramer method was used to adjust for multiple comparisons; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = 9.4, 95% CI 2-sided [5.0 to 13.7]

15. Secondary Outcome: Total Cholesterol Concentration
Description: Assessed from fasting blood draw expressed in mg/dL
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
mg/dL | 185 (1.69) | 193 (1.59)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Median Difference (Net) = -8.1, 95% CI 2-sided [-14.5 to -1.7]

16. Secondary Outcome: LDL Subclasses
Description: LDL subclasses with normal distribution; Measure Description: LDL particle size classifications are as follows: 22-25.5 nm is small, 25.6-26.5 nm medium, and 26.6-28.5 nm large. Typically, smaller LDL is associated with increased cardiovascular risk compared to larger.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
nmol/L
  Medium | 297 (20.2) | 337 (19.1)
  Small | 684 (24.5) | 677 (23.2)
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Results for medium subclass; Measure Description: LDL particle size classifications are as follows: 22-25.5 nm is small, 25.6-26.5 nm medium, and 26.6-28.5 nm large. Typically, smaller LDL is associated with increased cardiovascular risk compared to larger; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = -25.5, 95% CI 2-sided [-98.6 to 47.5]
Statistical Analysis 2: Comparison: Pecan Group vs Usual Care Group; Results for Small LDL particles; Measure Description: LDL particle size classifications are as follows: 22-25.5 nm is small, 25.6-26.5 nm medium, and 26.6-28.5 nm large. Typically, smaller LDL is associated with increased cardiovascular risk compared to larger; Test type: Superiority; Regression, Linear; adjustment for the baseline value, age (years), sex (male or female) and body mass index (BMI) (kg/m2); Mean Difference (Net) = 1.86, 95% CI 2-sided [-91.8 to 95.5]

17. Secondary Outcome: HDL Subclass-Large
Description: Measure was log transformed and back transformed to improve distribution; results for large HDL subclass are presented; Measure Description: Size classifications of HDL subclasses are as follows: large (size 9.4-14.0 nm), medium (8.3-9.3 nm), and small (7.3-8.2 nm). Higher levels of large HDL may be inversely related to cardiovascular risk.
Time Frame: 12 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Pecan Group | Usual Care Group
Number analyzed (Participants) | 62 | 68
μmol/L | 2.2 [2.0 to 2.3] | 2.0 [1.8 to 2.1]
Statistical Analysis 1: Comparison: Pecan Group vs Usual Care Group; Test type: Superiority; Regression, Linear; adjusted for outcome baseline value, age (years), sex (male or female) and baseline BMI (kg/m2); Mean Difference (Net) = 0.35, 95% CI 2-sided [0.07 to 0.63]

18. Other Pre Specified Outcome: Change in the Composition of the Gut Microbiota
Description: Abundance measured using 16 s rRNA sequencing
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: No deaths occurred no serious adverse events occurred.
Arm/Group | Pecan Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 2/69 | 0/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pecan Group (N=69) | Usual Care Group (N=69)
Appendectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant had appendectomy during the trial and was excluded from the remainder of the study
Gastric resection (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant underwent gastric resection during trial

LIMITATIONS AND CAVEATS:
Increased risk of type 1 statistical error. Dietary data was self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT05071807/Prot_004.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT05071807/SAP_005.pdf
  • Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT05071807/ICF_006.pdf